CLINICAL TRIAL: NCT04509310
Title: Effectiveness of Active Bodysuits for Adult Degenerative Scoliosis
Brief Title: Active Bodysuits for Adult Degenerative Scoliosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr. Kenny Kwan, Clinical Assistant Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW19-026; NCT03332277 (obsolete NCT alias)
Record Dates: First submitted 2020-06-05; First posted 2020-08-12 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Scoliosis
Keywords: Active Bodysuits
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active Bodysuits (Experimental): The potential materials that can provide support are 3D printable rigid materials, semirigid foam padding, Velcro tape and stretchable wide waistbands. The 3D printable materials can be very versatile in terms of properties and can be further finished with an epoxy resin or thermoplastics. Different compositions and structures of knitted fabrics will be used in different areas of the proposed bodysuits to provide a close fit, high breathability and effective pain management due to extra support. The fastening system includes a magnetic zipper and pulley system that can be adjusted by pulling on knobs. The pulley system contains a microadjustable dial, super-strong lightweight lacing, and low friction lacing guides.
  Interventions: Device: Active Bodysuits

INTERVENTIONS:
Device: Active Bodysuits — The wear trial period will be 9-12 months for each subject depending on the active biofeedback training progress. The bodysuits should provide active biofeedback training to the users. By incorporating the IMU sensors, the body alignment in the sagittal or coronal planes can be detected to provide feedback to the users via a wireless platform. This training will be customized to each individual user and will achieve a uniform body alignment goal that benefits the user. The participants will be assessed using the Scoliosis Research Society questionnaire (SRS-22r), the Oswestry Disability Index (ODI) and health-related quality-of-life (HRQOL) measures.

SUMMARY:
Adult degenerative (de novo) scoliosis (ADS) is a condition of the ageing population caused by degenerative changes without pre-existing spinal deformity. Pain is the most frequent problem, especially low back pain and radicular pain, and seriously affects the daily activities and health of ADS patients. The current treatment for ADS is not well defined. The main intervention for ADS treatment is surgical, but surgery is clearly not appropriate for every patient. Active bodysuits will be designed based on body alignment and pain management using special design components and incorporating active posture training from a biofeedback system. Back pain is often localized along the convexity of the curve, and passive support to the areas of pain, most likely in the lower trunk, hip and lower extremities, should be provided.

DETAILED DESCRIPTION:
The potential materials that can provide support are 3D printable rigid materials, semirigid foam padding, Velcro tape and stretchable wide waistbands. The 3D printable materials can be very versatile in terms of properties and can be further finished with an epoxy resin or thermoplastics. Different compositions and structures of knitted fabrics will be used in different areas of the proposed bodysuits to provide a close fit, high breathability and effective pain management due to extra support. The fastening system includes a magnetic zipper and pulley system that can be adjusted by pulling on knobs. The pulley system contains a microadjustable dial, super-strong lightweight lacing, and low friction lacing guides.

ELIGIBILITY:
Inclusion Criteria:

* Adults diagnosed with degenerative scoliosis
* Cobb's angle greater than 25 degrees
* Chronic lower back pain
* Limited mobility due to degenerative scoliosis

Exclusion Criteria:

* Substantial cardiac, pulmonary, renal or metabolic disease
* Neuromuscular scoliosis (e.g., spinal muscular atrophy, cerebral palsy, Parkinson's Disease, post-polio syndrome, Charcot Marie Tooth disease)
* Spine tumor, infection or connective tissue disorder
* Cognitively impaired or unable/unwilling to comply with follow-up
* Past history of vertebroplasty or kyphoplasty of the thoracic or lumbar spine

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-01-06 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Body alignment | 9-12 months
  Evaluation of kyphosis or lordosis in the sagittal plane

SECONDARY OUTCOMES:
Scoliosis Research Society Quality of Life Questionnaire | 1 year
  Scoliosis specific quality of life measure
Oswestry Disability Index | 1 year
  Back disability quality of life measure

CONTACTS AND LOCATIONS:
Overall Officials: Dr Kenny Kwan, BMBCh (Oxon), Principal Investigator — The University of Hong Kong
Locations (1):
- Duchess of Kent Children's Hospital, Hong Kong, Hong Kong